CLINICAL TRIAL: NCT06591819
Title: Safety of Hypofractionated Whole-Pelvis Proton Therapy With HDR Boost
Brief Title: Hypofractionated WPPT With HDR Boost
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 08824; 855972 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): The standard treatment for patients with prostate cancer is to receive brachytherapy boost and then radiation therapy in 25 fractions. This research study is being conducted to see how safe and effective delivering brachytherapy boost and then whole pelvis proton radiation therapy in 5 fractions (with each fraction having a higher dose than each fraction in the standard treatment) is in treating patients with prostate cancer. Subjects will also be asked to complete quality of life questionnaires for this study.
  Interventions: Radiation: Hypofractionated Whole Pelvis Proton Therapy with Brachytherapy Boost

INTERVENTIONS:
Radiation: Hypofractionated Whole Pelvis Proton Therapy with Brachytherapy Boost — Brachytherapy boost will be delivered and then whole pelvis proton radiation therapy in 5 fractions.

SUMMARY:
This is a phase II study of ultrahypofractionated whole pelvis proton therapy with brachytherapy boost for patients with high risk or unfavorable intermediate risk prostate with elevated risk of lymph node involvement.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic evidence of prostate cancer
* Risk group: high or intermediate risk as defined below

  * High risk: T3a or Gleason Grade Group 4/5 or PSA >20
  * Unfavorable intermediate risk disease: at least one or more of the following: T2b-T2c, Gleason Grade Group 2/3, PSA 10-20, >50% of cores positive
* Must be appropriate for whole pelvis per the treating oncologist or based on lymph node predicting nomogram
* Patient is a candidate for definitive external beam radiotherapy:

  * No prior radiotherapy in the region of study
  * No inflammatory bowel disease, active collagen/vascular/connective tissue disorders
* Age ³18 years
* ECOG performance status: 0-2
* Patients may initiate androgen deprivation therapy up to 3 months prior to radiation start, concurrently, or up to 3 months after completion of radiation therapy start. Patients may have received androgen deprivation therapy for the following months: unfavorable intermediate risk patients for 6 months; high-risk patients for 24 months. Patients will be allowed to discontinue ADT at physician and patient discretion.
* Pretreatment evaluation

  * History & Physical by a radiation oncologist within 6 weeks of enrollment
  * MRI prostate
  * PSMA PET
  * PSA level
* Eligible for rectal spacer procedure as determined by treating physician
* Informed consent: Patients must have the ability to understand and be willing to sign the study-specific informed consent indicating their understanding of the investigational nature and the risks of this study before any of the protocol related studies are performed (this does not include routine laboratory testing or imaging studies required to establish study eligibility);

Exclusion Criteria:

* Evidence of distant metastatic disease
* History of inflammatory bowel or active collagen/vascular/connective tissue disorders
* Prior radiation to the pelvis
* Prior or concurrent second invasive malignancy other than non-melanoma skin cancers, unless disease free for minimum of five years
* Known severe, active co-morbidity, defined as follows:

  o Any clinically significant unrelated systemic illness, medical condition, or other factor, which at the discretion of the Principal Investigators, would interfere in the safe and timely completion of study procedures, compromise the patient's ability to tolerate the protocol therapy, or is likely to interfere with the study procedures or results.
* Patients should not have a prior history of TURP
* Patients should not have pre-treatment IPSS >20 or on maximum alpha-blocker medications at baseline
* Patients should not be on therapeutic anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2034-01 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Safety of ultrahypofractionated proton therapy with HDR brachytherapy boost | First year of treatment
  The technique will be deemed safe if <10% of patients experience a CTCAE version 5.0 grade 3 or higher genitourinary or gastrointestinal toxicity cumulatively.

SECONDARY OUTCOMES:
Quality of life before and after radiotherapy | First year of treatment
  To evaluate for multiple domains of quality of life before and after radiotherapy by using validated surveys including EPIC-26 in urinary continence, urinary obstruction, bowel, and sexual domains. Investigators will determine minimally important differences for each domain.
Efficacy of proton radiotherapy | First year of treatment
  To determine treatment efficacy of proton radiotherapy for all enrolled patients as evidenced by biochemical control in the months following radiation. Investigators will follow PSA to determine if there is evidence for biochemical recurrence following radiotherapy. PSA recurrence will be defined as an increase of 2 ng/ml higher than the nadir value following completion of radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Goel, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No